CLINICAL TRIAL: NCT02960139
Title: A Pivotal, Prospective, Randomized, Controlled, Multicenter Superiority Clinical Study Comparing Standard Anastomosis Closure Technique to Standard Closure Technique Plus Sylys® Surgical Sealant
Brief Title: A Clinical Study Comparing Standard Anastomosis Closure Technique to Standard Closure Technique Plus Sylys® Surgical Sealant
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol updates resulted in new protocol/study
Sponsor: Cohera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO-106-0119
Record Dates: First submitted 2016-11-03; First posted 2016-11-09 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Colorectal and Ileorectal Anastomosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test- Treatment with Sylys Surgical Sealant (Experimental): Standard closure plus treatment with Sylys Surgical Sealant
  Interventions: Device: Test- Treatment with Sylys Surgical Sealan
- Control- Standard of Care (No Intervention): Control group is standard closure of anastomosis.

INTERVENTIONS:
Device: Test- Treatment with Sylys Surgical Sealan — Standard closure of stapled anastomosis plus treatment with Sylys Surgical Sealant
  Arms: Test- Treatment with Sylys Surgical Sealant

SUMMARY:
The Cohera Sylys® Surgical Sealant study is a pivotal, prospective, randomized, controlled, multicenter superiority clinical study comparing standard anastomosis closure technique (Control) to standard closure technique plus Sylys® Surgical Sealant (Test) during stapled colorectal and ileorectal anastomosis procedures.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 22 years of age
* Be scheduled for a stapled colorectal or ileorectal anastomosis procedure with or without diverting stoma
* Agree to return for all follow-up evaluations and procedures specified in the protocol
* Understand and give informed consent

Exclusion Criteria:

* Albumin < 3
* ASA ≥ 4
* Neutropenia ≤ 800
* Pregnancy
* The following conditions involving compromised immune system: AIDS (HIV positive not excluded), neutropenia
* Known blood clotting disorder requiring treatment
* Any condition known to effect wound healing, such as collagen vascular disease
* Have known or suspected allergy or sensitivity to any test materials or reagents
* Concurrent use of fibrin sealants or other anastomosis care devices
* Surgery for emergency abdominal indications
* Has undergone a colorectal anastomosis procedure in the previous two months
* Has an emergent infection related to a previous colorectal anastomosis procedure
* Is scheduled to undergo a Hartmann's procedure
* Is scheduled to undergo trans-anal endoscopic microsurgery (TEM) Is participating in another medical device trial related to colorectal anastomosis

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-04-13 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
A comparison of the incidence of anastomosis-related complications | from day of surgery to week 26

SECONDARY OUTCOMES:
A comparison of the proportion of patients who have incidence of sub-clinical or clinical anastomotic leaks | 14 days, 12 weeks, 26 weeks
  A comparison of the proportion of patients who have either sub-clinical or clinical anastomotic leaks in each group.

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - Flevoziekenhuis, Almere Stad, Flevoland
  - Meander Medical Center, Amersfoort
  - OLVG, Amsterdam
  - AMC, Amsterdam-Zuidoost
  - Laurentius, Roermond
  - Diakonessenhuis, Utrecht